CLINICAL TRIAL: NCT01380834
Title: Bilateral Paravertebral Blockade (T7-10) vs. Incisional Local Anesthetic Administration for Laparoscopic Cholecystectomy: a Prospective, Randomized Clinical Study
Brief Title: Bilateral Paravertebral Blockade (T7-10) vs. Incisional Local Anesthetic Administration for Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mihaela Visoiu (Other)
Responsible Party: Sponsor-Investigator, Mihaela Visoiu, Clinical Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO10060554; NCT01231048 (obsolete NCT alias)
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2015-05

CONDITIONS: Pain, Postoperative
Keywords: paravertebral nerve blocks; laparoscopic cholecystectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment group (Active Comparator): Group 1( treatment group ): 42 patients will have six paravertebral nerve blocks with ropivacaine 0.5 %, and incisional administration of placebo / normal saline at all four laparoscopic ports.
  Interventions: Drug: treatment group
- Placebo group (Placebo Comparator): Group 2(control group): 42 patients will have placebo/normal saline in paravertebral space, same amount, and injection at incision sites for all four insufflation ports with ropivacaine 0.5%.
  Interventions: Drug: control group

INTERVENTIONS:
Drug: control group — Group 2(control group): 42 patients will have placebo/normal saline in paravertebral space, same amount, and injection at incision sites for all four insufflation ports with ropivacaine 0.5%.
  Other Names: = Group 2(control group)
  Arms: Placebo group
Drug: treatment group — Group 1( treatment group ): 42 patients will have six paravertebral nerve blocks with ropivacaine 0.5 %, and incisional administration of placebo / normal saline at all four laparoscopic ports.
  Other Names: Group 1 ( treatment group)
  Arms: treatment group

SUMMARY:
The objective of this study is to assess the efficacy of paravertebral nerve blocks, single shot, with ropivacaine 0.5% for postoperative pain control after elective laparoscopic cholecystectomy as compared with incisional administration of same local anesthetic at laparoscopic insufflation ports by the surgeon.

DETAILED DESCRIPTION:
Pain after laparoscopic cholecystectomy is a result of many mechanisms such as tissue injury, local trauma to gallbladder removal, chemical irritation of the peritoneum, pneumoperitoneum. Effective analgesia in the immediate post-operative period following laparoscopic cholecystectomy is necessary for optimal recovery. Many methods for pain control after laparoscopic cholecystectomy have been evaluated, but none of them provided optimal postoperative analgesia. When used as a complement to general anesthesia, bilateral paravertebral blockade T5-T6 for adult laparoscopic cholecystectomy has been found to improve postoperative pain control. Whether this is also the case with pediatric patients is not certain. Analgesia from administration of local anesthetic by surgeon at insufflations ports is of short duration and may not provide sufficient pain relief. cholecystectomy.

84 pediatric patients (8-17 yrs old) will be randomly assigned to two groups: Group 1 (treatment group): 42 patients will have six paravertebral nerve blocks with ropivacaine 0.5%, and incisional administration of placebo / normal saline at all four laparoscopic ports.

Group 2 (control group): 42 patients will have placebo/normal saline in paravertebral space, same amount, and injection at incision sites for all for insufflation ports with ropivacaine 0.5%.

Both the anesthesiologist and the surgeon will be blinded to patient randomization.

Additional postoperative pain control will be provided via patient administered dilaudid PCA, for 12 hours after paravertebral block. After PCA is discontinued, the patient will receive oxycodone po and dilaudid iv for breakthrough pain.

Pain assessment will continue until 24 hours after paravertebral block or patient discharge if earlier than 24 hours.

The primary end-point of this research is the amount of dilaudid (ng/kg/min) administered via Patient Controlled Analgesia (PCA), 12 hours after administration of ropivacaine 0.5% /normal saline in paravertebral space and administration of normal saline/ropivacaine 0.5% at all four laparoscopic ports.

The secondary end points will be also for total amount of fentanyl (mcg/kg), dilaudid (mcg/kg), oxycodone (mg/kg) and morphine (mg/kg) (after conversion of above opioids to morphine based on opioids potency) used intraoperatively and 24 hours postoperatively (or until the patient is discharged, if sooner).

Postoperative pain scores will be assessed and compared at 4, 8, 12, 18 and 24 hr after paravertebral block using Visual Analog Scale (VAS).

Other secondary end-points will be possible side effects from opioids administration (nausea, emesis, itching, and episodes of respiratory depression) and possible complications associated with nerve blocks: pleural and vascular punctures, pneumothorax, back pain, bruises, and intravascular administration of local anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients scheduled for elective laparoscopic cholecystectomy under general anesthesia
* 8-17 yrs, female and male
* ASA 1, 2, 3
* more than 30 Kg
* BMI less than 36 (to calculate will use http://www.globalrph.com/bmi.htm )
* the patient must be able to self administer opioids via patient control analgesia (PCA)
* the patient must be able to complete postoperative questionnaires for pain score, pain type, location, patient satisfaction
* the patient will to be admitted for 24 hrs after surgery

Exclusion Criteria:

* patient refusal
* parental/guardian refusal
* history of coagulopathy, INR more than 1.5, platelets less than 100 000, PT , PTT more than normal value, patient on Coumadin, heparin or low molecular weight heparin ( LMWH)
* local infection at the planned block site
* vertebral anomalies, (e.g. scoliosis)
* BMI more or equal 36
* patient unable to self administer medications via PCA
* allergy to dilaudid, oxycodone, acetaminophen, ropivacaine
* chronic opioid use
* current weight less than 30 kg
* acute pain (pain on day of surgery that requires pain medication)
* pregnancy test positive

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2010-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Visoiu, MD, Principal Investigator — CHP of UPMC
Locations (1):
- Children's Hospital of Pittsburgh, UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Visoiu M, Cassara A, Yang CI. Bilateral Paravertebral Blockade (T7-10) Versus Incisional Local Anesthetic Administration for Pediatric Laparoscopic Cholecystectomy: A Prospective, Randomized Clinical Study. Anesth Analg. 2015 May;120(5):1106-1113. doi: 10.1213/ANE.0000000000000545. PMID 25427288

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group | Placebo Group
Started | 42 | 42
Completed | 41 | 42
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Placebo Group | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42 | 42 | 84
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14.5 [12 to 16] | 14 [12 to 15] | 14 [12 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 30 | 62
  Male | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Opioids Consumption Via PCA
Description: The primary end-point of this research is the amount of dilaudid (ng/kg/min) administered via Patient Controlled Analgesia (PCA), 12 hours after administration of ropivacaine 0.5% /normal saline in paravertebral space and administration of normal saline/ropivacaine 0.5% at all four laparoscopic ports.
Time Frame: 12 hrs after the blocks were done
Measure: Mean (Standard Deviation); unit: ng/kg/min
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 41 | 42
ng/kg/min | 107.29 (20.23) | 100.17 (46.77)

2. Secondary Outcome: Postoperative Pain Scores Assessed Using Visual Analog Scale (VAS).
Description: The VAS (Visual Analog Scale, 0 mm "no pain", to 100 mm," the worst pain possible ") is used to assess postoperative pain for patients. Postoperative pain scores will be assessed and compared at 4, 8, 12, 18 and 24 hr after paravertebral block.
Time Frame: 24 hrs after blocks were done or until the patient is discharged
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 41 | 42
units on a scale
  4h VAS | 42.68 (27.48) | 38.95 (26.94)
  8h VAS | 46.69 (30.15) | 37.67 (27.88)
  12h VAS | 43.88 (29.16) | 36.07 (27.94)
  18h VAS | 42.62 (31.22) | 35.73 (27.59)
  24h VAS | 42.17 (28.73) | 29.98 (25.91)

3. Secondary Outcome: Opioid Consumption
Description: Other secondary end points will total amount of fentanyl (mcg/kg), dilaudid (mcg/kg), oxycodone (mg/kg) and morphine (mg/kg) (after conversion of above opioids to morphine based on opioids potency) used at 24 hours postoperatively (or until the patient is discharged, if sooner).
Time Frame: 24 hrs after blocks were done or until the patient is discharged
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 41 | 42
mg/kg | 0.73 (0.32) | 0.71 (0.26)

ADVERSE EVENTS:
Arm/Group | Treatment Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/42
Other Adverse Events (participants affected / at risk) | 32/41 | 32/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=41) | Placebo Group (N=42)
Nausea (Gastrointestinal disorders) | 24 | 20
Emesis (Gastrointestinal disorders) | 14 | 15
Itching (Skin and subcutaneous tissue disorders) | 13 | 8
Back Pain (Injury, poisoning and procedural complications) | 3 | 1
Vascular Puncture (Injury, poisoning and procedural complications) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No